CLINICAL TRIAL: NCT03937921
Title: Dotarem Evaluation for Myocardial Perfusion CMR
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: Guerbet (Industry)
Responsible Party: Sponsor
Other Study IDs: 80969
Record Dates: First submitted 2019-04-17; First posted 2019-05-06 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Myocardial Perfusion Imaging; Magnetic Resonance Imaging
Keywords: Signal intensity enhancement; Relaxation rate enhancement
MeSH Terms: interventions — gadobutrol; Solutions; Injections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1 - Dotarem: Group 1 (n=30) will receive the clinically approved gadoterate meglumine (Dotarem, 0.1mmol/kg) as the contrast agent for their clinical perfusion study
- Group 2 - Gadavist: Group 2 (n=30) will receive the clinically approved gadobutrol (Gadavist, 0.1mmol/kg) as the contrast agent.
  Interventions: Drug: Gadavist 15Ml Solution for Injection

INTERVENTIONS:
Drug: Gadavist 15Ml Solution for Injection — Group 2 (n=30) will receive the clinically approved gadobutrol (Gadavist, 0.1mmol/kg) as contrast agent. The contrast agents will be administered at a flow rate of 5.0 ml/s for both groups. In this study aim, all imaging protocols will comply with standard of care and only the perfusion data will be post-processed and analyzed.
  Groups: Group 2 - Gadavist

SUMMARY:
The overall goal of this study is to investigate the signal intensity and relaxation rate characteristics of gadoterate meglumine (Dotarem, Guerbet, USA) enhanced myocardium during rest and stress perfusion cardiovascular magnetic resonance (CMR) compared to gadobutrol (Gadavist) to prove that Dotarem provides constantly high myocardial relaxation necessary for accurate quantitative perfusion evaluation.

The purpose of this study is to compare two types of contrast that patients receive during cardiac MRI scans to visualize the blood flow in the cardiac muscle. Both contrasts are used in standard of care procedures, and the one administered for each patient will be randomly selected. The length of the MRI study all procedures are the same as the clinically indicated scan.

DETAILED DESCRIPTION:
The overall goal of this study is to investigate the signal intensity and relaxation rate characteristics of gadoterate meglumine (Dotarem, Guerbet, USA) enhanced myocardium during rest and stress perfusion cardiovascular magnetic resonance (CMR) compared to gadobutrol (Gadavist) to prove that Dotarem provides constantly high myocardial relaxation necessary for accurate quantitative perfusion evaluation. Within this overall goal, the following specific aims will be pursued:

* Aim 1: To test the hypothesis that the signal intensity enhancement during Dotarem myocardial stress/rest perfusion is relatively constant, providing linear and stable enhancement in the myocardium, and is not inferior compared to gadobutrol (Gadavist).
* Aim 2: To test the hypothesis that the relaxation rate enhancement during Dotarem myocardial rest perfusion is uniform in the myocardium.

ELIGIBILITY:
Aim 1

Inclusion criteria:

To be eligible for the study: (All answers must be "YES" for subject to be eligible.)

1. Subject must be referred for a clinically indicated contrast-enhanced stress myocardial perfusion MRI scan out of concern of suspected myocardial ischemia.
2. Subject must be older than 18 years of age.
3. Subject must provide written informed consent prior to any study-related procedures being performed.
4. Subject must be willing to comply with all clinical study procedures.

Exclusion Criteria:

The presence of the following excludes subjects from the study: (All answers must be "NO" for subject to be eligible.)

1. Subject is a pregnant or nursing female. Exclude the possibility of pregnancy:

   * By testing (serum or urine beta HCG) within 24 hours before study date, or
   * By surgical sterilization, or
   * Post-menopausal, with minimum one (1) year history without menses.
2. Subject has an implanted cardiac pacemaker or implantable defibrillator.
3. Subject has a ferromagnetic vascular clip.
4. Subject has a neurostimulation system (e.g. TENS-Unit).
5. Subject has any type of cochlear implant.
6. Subject has ocular foreign body (e.g. metal shavings).
7. Subject carries any implanted device (e.g. insulin pump, drug infusion device).
8. Subject has shrapnel, bullet, or other type of metal fragments within the body.
9. Subject has an acute psychiatric disorder or is cognitively impaired.
10. Subject is using or is dependent on substances of abuse.
11. Subject is unwilling to comply with the requirements of the protocol.
12. Subject is in acute unstable condition.
13. Subject has an allergy against gadolinium based contrast agents or pharmaceutical stressors used in this study.
14. Subject has impaired renal function (creatinine > 1.5 mg/dl).
15. Subject presenting with acute coronary syndrome.
16. Positive cardiac enzymes positive troponin, CK-MB, or myosin
17. ST-elevations, new transient ST changes greater than 0.05mV or T- wave inversions with symptoms

Aim 2

Inclusion criteria:

To be eligible for the study: (All answers must be "YES" for subject to be eligible.)

1. Subject must be referred for a clinically indicated contrast-enhanced stress myocardial perfusion MRI scan out of concern of suspected myocardial ischemia.
2. Subject must be older than 18 years of age.
3. Subject must provide written informed consent prior to any study-related procedures being performed.
4. Subject must be willing to comply with all clinical study procedures.

Exclusion Criteria:

The presence of the following excludes subjects from the study: (All answers must be "NO" for subject to be eligible.)

1. Subject is a pregnant or nursing female. Exclude the possibility of pregnancy:

   * By testing (serum or urine beta HCG) within 24 hours before study date, or
   * By surgical sterilization, or
   * Post-menopausal, with minimum one (1) year history without menses.
2. Subject has an implanted cardiac pacemaker or implantable defibrillator.
3. Subject has a ferromagnetic vascular clip.
4. Subject has a neurostimulation system (e.g. TENS-Unit).
5. Subject has any type of cochlear implant.
6. Subject has ocular foreign body (e.g. metal shavings).
7. Subject carries any implanted device (e.g. insulin pump, drug infusion device).
8. Subject has shrapnel, bullet, or other type of metal fragments within the body.
9. Subject has an acute psychiatric disorder or is cognitively impaired.
10. Subject is using or is dependent on substances of abuse.
11. Subject is unwilling to comply with the requirements of the protocol.
12. Subject is in acute unstable condition.
13. Subject has an allergy against gadolinium based contrast agents used in this study.
14. Subject has impaired renal function (creatinine > 1.5 mg/dl).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There will not be any eligibility criteria for any subpopulations. In addition, there will not be any targeted involvement of special classes of subjects, such as fetuses, neonates, pregnant women, children, prisoners, institutionalized individuals, or others who may be considered vulnerable populations. All race and ethnicities and both genders will be considered for inclusion into the study. Subjects under the age of 18 will not be considered for inclusion into this study.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2019-07-03 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Signal intensity of gadoterate meglumine during perfusion cardiovascular magnetic resonance | 1 year
  Characteristics of signal intensity changes and absolute myocardial blood flow using the MASS Research Software; signal intensity-time curves from the perfusion data

SECONDARY OUTCOMES:
Relaxation rate characteristics of gadoterate meglumine during perfusion cardiovascular magnetic resonance | 1 year
  The uniformity of T1 and R1 (inverse T1) evaluated using the MASS Research Software; equilibrium T1 maps generated by pre-contrast T1 and repeat inversion recovery images during the perfusion of the coronary arteries

CONTACTS AND LOCATIONS:
Overall Officials: Joseph U. Schoepf, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT03937921/Prot_SAP_000.pdf
  • Informed Consent Form (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/21/NCT03937921/ICF_001.pdf